CLINICAL TRIAL: NCT03328520
Title: WILD 5 Wellness, A 30 Day Intervention in First Year Students at Beloit College
Brief Title: WILD 5 Wellness, A 30-Day Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beloit College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 374
Record Dates: First submitted 2017-10-20; First posted 2017-11-01 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Depression; Cognitive Functioning; Wellness
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First Year Students in Wellness FYIs (Experimental)
  Interventions: Behavioral: WILD 5 Wellness Intervention

INTERVENTIONS:
Behavioral: WILD 5 Wellness Intervention — Behaviors in 6 areas of wellness: Sleep, Social Connectedness, Exercise, Nutrition, Mindfulness and "HERO" (Happiness, Enthusiasm, Resilience, Optimism)

SUMMARY:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition in First Year Beloit College students self-selected into a wellness focused first year initiative. This program is called "WILD 5 Wellness: A 30-Day Intervention".

ELIGIBILITY:
Inclusion Criteria:

* Students 18 years of age or older or 17 years of age with legal guardian written permission.
* Students enrolled in First Year Initiative Courses titled "Balance" or "Constructing Health"

Exclusion Criteria:

* Individuals who are pregnant or plan to get pregnant during the next 30 days.
* Students who are not enrolled in the First Year Initiative Courses titled "Balance" or "Constructing Health"

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Day 0, Day 30+ 3 days (approximately)
  PHQ-9 is a self reported depression scale. It is a 9-item scale with scores ranging from 0-27. Lower scores denote improvement.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Day 0, Day 30+ 3 days (approximately)
  GAD-7 is a self-reported questionnaire used to assess anxiety symptoms. It is a 7-item scale with scores ranging from 0-21. Lower score denotes improvement.
Change in the HERO Wellness Scale | Day 0, Day 30+ 3 days (approximately)
  HERO Wellness Scale is a brief scale designed to measure mental wellness specifically happiness, enthusiasm, resilience and optimism. It is a 5-item scale with scores ranging from 0-10. Higher score denotes improvement.
Change in World Health Organization-5 (WHO-5) | Day 0, Day 30+ 3 days (approximately)
  WHO-5 is a brief scale that measures mental well-being. It is a 5-item scale with scores ranging from 0-25. Higher score denotes improvement.
Change in Cognitive and Physical Functioning Questionnaire (CPFQ) | Day 0, Day 30+ 3 days (approximately)
  CPFQ is a brief scale that measures cognitive and executive dysfunction. It is a 7-item scale with scores ranging from 7-42. Lower score denotes improvement.

SECONDARY OUTCOMES:
The Post-Program Participant Questionnaire | Day 30+ 3 days (approximately)
  The Post-Program Participant Questionnaire is a brief survey that captures participants'opinions about WILD 5 Wellness.

CONTACTS AND LOCATIONS:
Overall Officials: Tara M Girard, BSN, Principal Investigator — Beloit College; Suzanne Cox, PhD, Principal Investigator — Beloit College; Laura Parmentier, PhD, Principal Investigator — Beloit College; Saundra Jain, PsyD, LPC, Principal Investigator — Beloit College; Rakesh Jain, MD, MPH, Principal Investigator — Beloit College
Locations (1):
- Beloit College, Beloit, Wisconsin, United States